CLINICAL TRIAL: NCT00804752
Title: Vitamin D Treatment in Patients With Chronic Hepatitis C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Dr. Saif Abu-Mouch, Hepatology Clinic, Hillel Yaffe Medical Center
Other Study IDs: 0040-08-HYMC
Record Dates: First submitted 2008-12-07; First posted 2008-12-09 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Chronic Hepatitis C
Keywords: Patients with Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Vitamin D

ARMS (1):
- Vitamin D (Experimental): An addition of Vitamin D to the standard treatment
  Interventions: Drug: Adding vitamin D; Drug: Vitamin D

INTERVENTIONS:
Drug: Adding vitamin D — Adding 1000IU/Vitamin D daily
Drug: Vitamin D — Addition of 1000IU/day Vitamin D

SUMMARY:
We hypothesize that patients with Ch.HCV have a low level of vitamin D, and that by raising their vitamin D levels by adding it to their standard treament of Pegylated Interferon and Ribavirin, there will be an increase in their sustained virological response.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hepatitis C Genotype 1

Exclusion Criteria:

* Vitamin D intoxication Renal Failure Liver Failure Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
To increase the sustained virological response | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel